CLINICAL TRIAL: NCT00690599
Title: Socioeconomic Profile and Patient Satisfaction Assessment in an Academic Dental General Clinic
Brief Title: Socioeconomic Profile and Patient Satisfaction Assessment
Acronym: Satisfaction
Status: Completed | Type: Observational
Sponsor: Fortaleza University (Other)
Responsible Party: Carlos Antonio Bruno da Silva/ Phd, Universidade de Fortaleza
Other Study IDs: 07-125
Record Dates: First submitted 2008-05-30; First posted 2008-06-04 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-05

CONDITIONS: Satisfaction; Dentist-Patient Relations
Keywords: Patient satisfaction; Dentist-Patient relations; Answering services
MeSH Terms: conditions — Personal Satisfaction; Patient Satisfaction

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the study was to evaluate the socioeconomic patient's profile and their level of satisfaction in the general dental practice clinic. A cross-sectional quantitative study was accomplished with 80 patients assisted at the referred service. A solely-applied questionnaire was used regarding the following aspects: structure and environment, fear and anxiety, reliability, empathy and commitment, resolutivity and quality of the accomplished services. It was observed that the assisted patients' profile consisted predominantly of a female sample (71,2%), that completed the medium learning (31,2%) and/or that didn't finish the fundamental level (26,2%). Moreover 50% of them presented a family income of 1 to 2 minimum salaries and 41,2% were unemployed. As the quality of the rendered technical service, nearly 70% of the users considered it great, as well as the clinic's structure and environment. Regarding the satisfaction with to the received treatment, 76,2% of the interviewees gave the maximum score of 10 and 95% would recommend the attendance to others. It is concluded that the patients are satisfied with the clinical attendance accomplished by the students in the general practice dental clinic at UNIFOR, in what refers to its technical and functional quality.

ELIGIBILITY:
Inclusion Criteria:

* Patient registered in Academic of Information System (SIA),
* Patient assisted in the general dental clinic,
* To have 18 years or more or to be parents accompanied,
* Agree with research participation.

Exclusion Criteria:

* To be urgency patient,
* To be the first day of attendance at clinic.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients assisted in the general dental practice clinic at UNIFOR Ceará - Brazil.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2006-04; Primary Completion 2006-05 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Solange K Saito, PhD, Principal Investigator — Fortaleza University
Locations (1):
- Fortaleza University, Fortaleza, Ceará, Brazil

REFERENCES:
- See also: Fortaleza University — http://www.unifor.br